CLINICAL TRIAL: NCT02557295
Title: An Observational, Prospective Cohort Study to Evaluate Safety and Efficacy of Remsima™ in Patients With Rheumatoid Arthritis
Brief Title: An Observational Study to Evaluate Safety and Efficacy of Remsima™ in Patients With RA
Status: Terminated | Type: Observational
Why Stopped: Terminated
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-P13 4.2
Record Dates: First submitted 2015-03-18; First posted 2015-09-23 (Estimated); Results first posted 2024-02-05 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Remsima™: Patients who have received only Remsima or switched from non-biologic treatment to Remsima were included in this analysis group.
- Switch to Remsima I: Patients who switched from Remicade to Remsima were included in this analysis group.
- Switch to Remsima II: Patients who switched to Remsima from biologic treatment other than Remicade were included in this analysis group.
- Remicade: Patients who have received only Remicade or switched from non-biologic treatment to Remsima were included in this analysis group.
- Switch to Remicade I: Patients who switched from Remsima to Remicade were included in this analysis group.
- Switch to Remicade II: Patients who switched to Remicade from biologic treatment other than Remsima will be included in this analysis group.
- Other Anti-TNF: Following patients were included in other anti-TNF group.
  * Patients who have received only anti-TNF other than Remsima or Remicade
  * Patients who switched from non-biologic treatment to anti-TNF other than Remsima or Remicade
  * Patients who switched from biologic treatment other than anti-TNF before study enrolment to anti-TNF other than Remsima or Remicade
- Switch to Other Anti-TNF: Patients who switched from Remsima or Remicade to other anti-TNF other than Remicade will be included in this analysis group
- Biologic Naïve: Patients who received only non-biologic treatment will be included in this analysis group

SUMMARY:
An Observational, Prospective Cohort Study to Evaluate Safety and Efficacy of RemsimaTM in Patients with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This is a longitudinal, observational, prospective cohort study to assess the safety and efficacy of RemsimaTM in patients with RA in comparison with patients receiving non-biologic treatmentsor other anti-TNF drugs. For the RemsimaTM cohort data will be collected for patients who commence treatment with RemsimaTM in accordance with the product label at the time of enrolment (3 mg/kg of RemsimaTM by IV infusion at weeks 0, 2, 6 (±3 days) and every 8 weeks (±14 days) thereafter). For patients who have been treated with Remicade® prior to enrolment, their dosing schedule will be continued appropriately. This observational study allows drug switching between anti-TNF drugs. If switched to RemsimaTM, data will be collected until the end of study for each patient. If switched to other anti-TNF drugs (infliximab (Remicade®), etanercept, adalimumab and etc.), data will be collected until 1 year from the day of switch or until the end of study for each patient, whichever reaches earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Patients with active RA diagnosed according to the revised 1987 ACR or 2010 ACR/EULAR classification criteria

Exclusion Criteria:

1. Patients with a history of hypersensitivity to murine, chimeric, human, or humanized proteins.
2. Patients with a current or past history of chronic infection
3. Patients with moderate or severe heart failure (NYHA class III/IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of at least 950 male and female patients with Rheumatoid Arthritis
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2013-12-17 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klara Sirova, Principal Investigator — Revmatologie MUDr. Klara Sirova s.r.o. Chelčického 616/12 , 702 00, Czech Republic

REFERENCES:
- [Derived] Cheon JH, Nah S, Kang HW, Lim YJ, Lee SH, Lee SJ, Kim SH, Jung NH, Park JE, Lee YJ, Jeon DB, Lee YM, Kim JM, Park SH. Infliximab Biosimilar CT-P13 Observational Studies for Rheumatoid Arthritis, Inflammatory Bowel Diseases, and Ankylosing Spondylitis: Pooled Analysis of Long-Term Safety and Effectiveness. Adv Ther. 2021 Aug;38(8):4366-4387. doi: 10.1007/s12325-021-01834-3. Epub 2021 Jul 12. PMID 34250583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant flow was summarized by all analysis groups as prespecified in Statistical Analysis Plan.
  According to study protocol inclusion criteria, without prior RA medication restrictions, patients who received Remsima, Remicade, Other anti-TNF and biologic naïve were enrolled and switching between were allowed
Pre-assignment Details: A total of 302 patients were screened, and 248 patients were enrolled.
Groups:
- Remsima: Patients who have received only Remsima or switched from non-biologic treatment to Remsima were included in this analysis group.
- Switch to Remsima: Patients who switched from Remicade to Remsima were included in this analysis group.
- Remicade: Patients who have received only Remicade or switched from non-biologic treatment to Remicade were included in this analysis group.
- Switch to Remicade: Patients who switched from Remsima to Remicade were included in this analysis group.
Period: Overall Study
Arm/Group | Remsima | Switch to Remsima | Switch to Remsima II | Remicade | Switch to Remicade | Switch to Remicade II | Other Anti-TNF | Switch to Other Anti-TNF | Biologic Naïve
Started | 111 | 8 | 15 | 3 | 0 | 0 | 81 | 7 | 23
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 111 | 8 | 15 | 3 | 0 | 0 | 81 | 7 | 23
Not completed — Withdrawal by Subject | 9 | 2 | 4 | 0 | 0 | 0 | 15 | 1 | 3
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 24 | 1 | 3 | 0 | 0 | 0 | 12 | 1 | 0
Not completed — Adverse Event | 16 | 2 | 3 | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
Not completed — Study Close | 54 | 3 | 5 | 3 | 0 | 0 | 37 | 3 | 19
Not completed — except for study close | 4 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients data were analyzed; however, there were 0 patients recruited in the "Switch to Remicade I" and "Switch to Remicade II" groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Remsima | Switch to Remsima I | Switch to Remsima II | Remicade | Switch to Remicade I | Switch to Remicade II | Other Anti-TNF | Switch to Other Anti-TNF | Biologic Naïve | Total
Number analyzed (Participants) | 111 | 8 | 15 | 3 | 0 | 0 | 81 | 7 | 23 | 248
Age, Continuous [Median (Full Range); unit: years] | 55.0 [27 to 78] | 57.5 [48 to 71] | 56 [27 to 67] | 53.0 [52 to 56] |  |  | 53.0 [22 to 75] | 44 [29 to 58] | 54 [38 to 78] | 54.6 [22 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 7 | 13 | 1 |  |  | 65 | 6 | 22 | 198
  Male | 27 | 1 | 2 | 2 |  |  | 16 | 1 | 1 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0
  Asian | 98 | 8 | 13 | 3 |  |  | 74 | 7 | 23 | 226
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0
  White | 13 | 0 | 2 | 0 |  |  | 7 | 0 | 0 | 22
  More than one race | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number and Percentage of Patients With the Following Adverse of Events of Special Interest (ESI)
Description: * Hepatitis B virus reactivation
  * Congestive heart failure
  * Opportunistic infections (excluding tuberculosis)
  * Serious infections including sepsis (excluding opportunistic infections and tuberculosis)
  * Tuberculosis (TB)
  * Serum sickness (delayed hypersensitivity reactions)
  * Haematological reactions
  * Systemic lupus erythematosus/lupus-like syndrome
  * Demyelinating disorders
  * Lymphoma (not hepatosplenic T cell lymphoma)
  * Hepatobiliary events
  * Hepatosplenic T cell lymphoma (HSTCL)
  * Serious infusion reactions during a re-induction regimen following disease flare
  * Sarcoidosis/sarcoid-like reactions
  * Leukaemia
  * Malignancy (excluding lymphoma)
  * Skin cancer
  * Pregnancy exposure
  * Infusion reactions associated with shortened infusion duration
  * Infusion related reaction (IRR)/hypersensitivity/anaphylactic reaction
Time Frame: Duration of study participation (up to 5 years)
Population: The analysis period for patients with one switching after enrollment were defined as the whole period beginning on the date of first switching, for patients with two or more switching after enrollment, the period between first and second switching was used. All patients data were analyzed; however, there were 0 patients recruited in the "Switch to Remicade I" and "Switch to Remicade II" groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Remsima | Switch to Remsima I | Switch to Remsima II | Remicade | Switch to Remicade I | Switch to Remicade II | Other Anti-TNF | Switch to Other Anti-TNF | Biologic Naïve
Number analyzed (Participants) | 111 | 8 | 15 | 3 | 0 | 0 | 81 | 7 | 23
Participants
  TEAE of Serious infections including sepsis (excluding opportunistic infections and tuberculosis) | 5 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  TEAE of tuberculosis | 7 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  TEAE of Haematological reactions | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  TEAE of Systemic lupus erythematosus/lupus-like syndrom | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE of Hepatobiliary events | 6 | 1 | 1 | 1 | 0 | 0 | 5 | 0 | 1
  TEAE of Malignancies (excluding lymphoma) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  TEAE of Infusion reactions associated with shortened infusion duration | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE of Infusion related reaction/hypersensitivity/ anaphylactic reaction | 15 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 0

2. Secondary Outcome: Descriptive Statistics of Disease Activity Score in 28 Joints (DAS28) (ESR) and DAS28 (CRP)
Description: Disease activity score in 28 joints (DAS28) will be calculated in two ways using the following two equations: DAS28(ESR) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.70 × ln(ESR)) + (0.014 × GH); DAS28(CRP) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.36 × ln(CRP + 1)) + (0.014 × GH) + 0.96
  Where:
  TJC28 = number of tender joints (0-28): tender joint count (TJC); SJC28 = number of swollen joints (0-28): swollen joint count (SJC); ESR = ESR measurement (mm/h); CRP = CRP measurement (mg/L); GH = Patient Global Assessment of Disease Activity measured on VAS (0 - 100 mm)
  Disease activity is indexed as follows, on a 10 point scale, with higher numbers indicating worse disease activity:
  Remission: DAS28 < 2.6 Low Disease Activity: 2.6 ≤ DAS28 < 3.2 Moderate Disease Activity: 3.2 ≤ DAS28 ≤ 5.1 High Disease Activity: 5.1 < DAS28
Time Frame: Day 0 ~ Week 198 (every 6 months ±6 weeks)
Population: The Efficacy Analysis set consisted of all patients who received at least one infliximab dose (Remsima or Remicade) and providing at least one post treatment efficacy result during analysis period. Efficacy analysis was only performed in the Remsima, Switch to Remsima, Remicade and Switch to Remicade analysis groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remsima | Switch to Remsima | Remicade | Switch to Remicade
Number analyzed (Participants) | 80 | 3 | 3 | 0
score on a scale
  Day 0 DAS28 (ESR): number analyzed (Participants) | 71 | 3 | 2 | 0
  Day 0 DAS28 (ESR) | 5.698 (1.1035) | 4.212 (1.6056) | 5.195 (0.8118) |
  Week 30 DAS28 (ESR): number analyzed (Participants) | 66 | 3 | 3 | 0
  Week 30 DAS28 (ESR) | 3.575 (1.4181) | 3.833 (1.5004) | 3.509 (2.2685) |
  Week 54 DAS28 (ESR): number analyzed (Participants) | 37 | 3 | 1 | 0
  Week 54 DAS28 (ESR) | 3.574 (1.3803) | 3.877 (1.3921) | 1.456 |
  Week 78 DAS28 (ESR): number analyzed (Participants) | 14 | 0 | 1 | 0
  Week 78 DAS28 (ESR) | 3.028 (1.2306) |  | 1.282 |
  Week 102 DAS28 (ESR): number analyzed (Participants) | 6 | 0 | 0 | 0
  Week 102 DAS28 (ESR) | 2.780 (0.7859) |  |  |
  Week 126 DAS28 (ESR): number analyzed (Participants) | 3 | 0 | 0 | 0
  Week 126 DAS28 (ESR) | 2.573 (0.6413) |  |  |
  Week 150 DAS28 (ESR): number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 150 DAS28 (ESR) | 2.300 |  |  |
  Week 174 DAS28 (ESR): number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 174 DAS28 (ESR) | 2.090 |  |  |
  Week 198 DAS28 (ESR): number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 198 DAS28 (ESR) | 3.100 |  |  |
  Day 0 DAS28 (CRP): number analyzed (Participants) | 67 | 3 | 2 | 0
  Day 0 DAS28 (CRP) | 5.016 (1.1541) | 3.172 (2.0141) | 4.763 (0.9537) |
  Week 30 DAS28 (CRP): number analyzed (Participants) | 65 | 3 | 3 | 0
  Week 30 DAS28 (CRP) | 2.969 (1.2336) | 2.775 (1.3919) | 3.665 (1.7950) |
  Week 54 DAS28 (CRP): number analyzed (Participants) | 38 | 3 | 1 | 0
  Week 54 DAS28 (CRP) | 2.963 (1.3779) | 2.854 (1.3705) | 1.172 |
  Week 78 DAS28 (CRP): number analyzed (Participants) | 14 | 0 | 1 | 0
  Week 78 DAS28 (CRP) | 2.583 (1.0857) |  | 1.219 |
  Week 102 DAS28 (CRP): number analyzed (Participants) | 6 | 0 | 0 | 0
  Week 102 DAS28 (CRP) | 1.979 (0.7980) |  |  |
  Week 126 DAS28 (CRP): number analyzed (Participants) | 3 | 0 | 0 | 0
  Week 126 DAS28 (CRP) | 2.200 (0.7632) |  |  |
  Week 150 DAS28 (CRP): number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 150 DAS28 (CRP) | 2.050 |  |  |
  Week 174 DAS28 (CRP): number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 174 DAS28 (CRP) | 2.720 |  |  |
  Week 198 DAS28 (CRP): number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 198 DAS28 (CRP) | 2.680 |  |  |

3. Secondary Outcome: Descriptive Statistics for Actual Value of Health Assessment Questionnaire (HAQ) Estimate of Physical Ability
Description: The arthritis-related functional disability will be measured using the disability index of the Health Assessment Questionnaire (HAQ), a validated, self-administered form that assesses functional ability in a number of relevant areas, including the ability to dress, rise from bed, eat, walk, maintain personal hygiene, reach, grip and other activities on a scale ranging from 0 (without any difficulty) to 3 (unable to do). Scores range from 0 to 3, with higher scores indicating worse disability.
  There are 8 categories within the Health Assessment Questionnaire. The answer to each question will be scored as follows: Without any difficulty = 0, With some difficulty = 1, With much difficulty = 2, Unable to do = 3.
  Divide the summed category scores (using the adjustment score) by the number of categories answered to obtain the HAQ estimate of physical ability.
Time Frame: Day 0 ~ Week 198 (every 6 months ±6 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remsima | Switch to Remsima | Remicade | Switch to Remicade
Number analyzed (Participants) | 80 | 3 | 3 | 0
score on a scale
  Day 0 HAQ: number analyzed (Participants) | 73 | 3 | 2 | 0
  Day 0 HAQ | 1.0377 (0.64472) | 0.5417 (0.83229) | 1.1875 (1.14905) |
  Week 30 HAQ: number analyzed (Participants) | 69 | 3 | 3 | 0
  Week 30 HAQ | 0.6141 (0.60167) | 0.5000 (0.50000) | 0.7500 (1.08972) |
  Week 54 HAQ: number analyzed (Participants) | 42 | 3 | 3 | 0
  Week 54 HAQ | 0.7173 (0.69955) | 0.3333 (0.47324) | 0.4583 (0.59073) |
  Week 78 HAQ: number analyzed (Participants) | 20 | 0 | 1 | 0
  Week 78 HAQ | 0.6813 (0.63670) |  | 0.0000 |
  Week 102 HAQ: number analyzed (Participants) | 11 | 0 | 0 | 0
  Week 102 HAQ | 0.6364 (0.52278) |  |  |
  Week 126 HAQ: number analyzed (Participants) | 3 | 0 | 0 | 0
  Week 126 HAQ | 0.2917 (0.40182) |  |  |
  Week 150 HAQ: number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 150 HAQ | 0.1250 |  |  |
  Week 174 HAQ: number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 174 HAQ | 0.0000 |  |  |
  Week 198 HAQ: number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 198 HAQ | 0.6250 |  |  |

ADVERSE EVENTS:
Time Frame: Duration of study participation (up to 5 years)
Description: The analysis period for patients with one switching after enrollment were defined as the whole period beginning on the date of first switching, for patients with two or more switching after enrollment, the period between first and second switching was used.
Arm/Group | Remsima | Switch to Remsima I | Switch to Remsima II | Remicade | Switch to Remicade I | Switch to Remicade II | Other Anti-TNF | Switch to Other Anti-TNF | Biologic Naïve
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/8 | 0/15 | 0/3 | 0/0 | 0/0 | 0/81 | 0/7 | 0/23
Serious Adverse Events (participants affected / at risk) | 16/111 | 2/8 | 4/15 | 2/3 | 0/0 | 0/0 | 11/81 | 0/7 | 2/23
Other Adverse Events (participants affected / at risk) | 56/111 | 6/8 | 7/15 | 3/3 | 0/0 | 0/0 | 39/81 | 3/7 | 13/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remsima (N=111) | Switch to Remsima I (N=8) | Switch to Remsima II (N=15) | Remicade (N=3) | Switch to Remicade I (N=0) | Switch to Remicade II (N=0) | Other Anti-TNF (N=81) | Switch to Other Anti-TNF (N=7) | Biologic Naïve (N=23)
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remsima (N=111) | Switch to Remsima I (N=8) | Switch to Remsima II (N=15) | Remicade (N=3) | Switch to Remicade I (N=0) | Switch to Remicade II (N=0) | Other Anti-TNF (N=81) | Switch to Other Anti-TNF (N=7) | Biologic Naïve (N=23)
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic Cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis Acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 13 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Latent Tuberculosis (Infections and infestations) | 7 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Nasopharyngitis (Infections and infestations) | 10 | 1 | 1 | 0 | 0 | 0 | 7 | 1 | 0
Tinea Pedis (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 0 | 1 | 0 | 0 | 0 | 12 | 0 | 0
Vaginal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Lactation Disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localized Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menopausal disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dydspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-06-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT02557295/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT02557295/SAP_001.pdf